CLINICAL TRIAL: NCT05074251
Title: Pilot Study of Secondary Distribution of HIV Self-screening Tests by Women With HIV: An Innovative Strategy to Improve Testing, Identification, and Linkage to Treatment of Men in South Africa
Brief Title: Evaluation of Secondary Distribution of HIV Self-screening Tests by Women With HIV
Acronym: HIVSSSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Emory University (Other); BroadReach Healthcare (Industry); United States Agency for International Development (USAID) (U.S. Federal Agency); Mpumalanga Department of Health (Other Government)
Responsible Party: Principal Investigator, Dvora Joseph Davey, PhD, MPH, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRHIVSTSA1
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Results first posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-03

CONDITIONS: HIV Infections; ART; HIV Seropositivity
Keywords: HIV self testing; HIV self screening; South Africa
MeSH Terms: conditions — HIV Infections; HIV Seropositivity | interventions — Counseling; Referral and Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIV self testing (Experimental): HIV+ women will receive HIV self-tests (2) to bring home to her partner to offer for testing
  Interventions: Diagnostic Test: HIV self test; Behavioral: Counseling and referral for partner testing
- Standard of care (Active Comparator): In the standard of care arm, women will receive standard of care partner referrals for HIV testing, including counselling about disclosure and referral for her partner(s) to return to the facility for testing.
  Interventions: Behavioral: Counseling and referral for partner testing

INTERVENTIONS:
Diagnostic Test: HIV self test — For women allocated to the intervention arm, the participant will be given HIV self testing and counseling on their use & importance of partner testing, to take home to their partner(s).
  Other Names: counseling on partner testing and HIV self testing
  Arms: HIV self testing
Behavioral: Counseling and referral for partner testing — Counseling and refer participant's partner for facility based HIV testing

SUMMARY:
Many South African men do not visit clinics or get tested due to multiple real and perceived barriers. Nkangala District has significant gaps to identifying PLHIV who are not on ART, reaching their ART targets, especially in adult men. Over 65% of PLHIV not on ART are men, which is a gap of over 39,000 men living with HIV needing to be tested and initiated on ART.

* To improve case finding among men in Nkangala we will evaluate how best to reach partners of PLHIV (newly diagnosed or on ART) with index testing by using HIV self-screening (HIVSS) and linkage to ART start.
* Secondary distribution of HIV self-screening kits (HIVSS), whereby clients bring HIVSS kits to their partners, addresses barriers by enabling partners to screen themselves at their convenience and in the privacy of their homes.

Study Objectives: BroadReach in collaboration with UCLA, UCT and Nkangala DOH will pilot test an innovative index partner HIVSS strategy in one urban and one rural clinic to evaluate acceptability, barriers, and efficacy of secondary HIVSS distribution in a randomized control trial enrolling women newly diagnosed with HIV or on ART.

* In the intervention arm, women will receive counselling on how to use HIVSS, how to encourage their male partner to screen, and 2 oraquick HIVSS with instructions and invitation to return for confirmatory testing.
* In the standard of care arm, index women will receive counselling on the importance of disclosure to their family and partner(s) and referral for HIV testing (per South African national guidelines).

Study design: Randomized control trial of n=180 WLHIV (90 in each arm) in four facilities (urban and rural) in the Nkangala district ensure that the results are generalizable.

DETAILED DESCRIPTION:
Many South African men do not visit clinics or get tested due to multiple real and perceived barriers. Nkangala District has significant gaps to identifying PLHIV who are not on ART, reaching their ART targets, especially in adult men. Over 65% of PLHIV not on ART are men, which is a gap of over 39,000 men living with HIV needing to be tested and initiated on ART.

* To improve case finding among men in Nkangala we will evaluate how best to reach partners of PLHIV (newly diagnosed or on ART) with index testing by using HIV self-screening (HIVSS) and linkage to ART start.
* Secondary distribution of HIV self-screening kits (HIVSS), whereby clients bring HIVSS kits to their partners, addresses barriers by enabling partners to screen themselves at their convenience and in the privacy of their homes.

We will partner with BroadReach Healthcare, a PEPFAR partner in South Africa, to pilot test an innovative index partner HIVSS strategy in one urban and one rural public health clinic in the Nkangala district of Mpumalanga Province to evaluate acceptability, barriers, and preliminary efficacy of secondary HIVSS distribution in a randomized control trial enrolling women newly diagnosed with HIV or on ART. In the intervention arm, women will receive counselling on how to use HIVSS, how to encourage their male partner to screen, and 2 HIVSSs with HIVSS instructions and invitation to return for confirmatory testing. In the standard of care arm, index women will receive counselling on the importance of disclosure to their family and partner(s) and referral for HIV testing (per SA national guidelines). We will evaluate the following aims:

1. Conduct a mixed-methods survey with N=180 HIV+ women to assess perceived acceptability and barriers (including perceived safety, IPV) to secondary HIVSS distribution by women to male partners.
2. Test the feasibility and preliminary efficacy of secondary HIVSS distribution through a 1:1 randomized control trial in n=180 HIV+ women to assess, comparing standard of care to intervention arm:

   1. % of index women who self-report that they gave the HIVSS or standard of care referral for testing to their male partner
   2. % of male partners who either screened or tested for HIV assessed at 3 months after randomization (primary outcome)

   i. Measured via options of: index or partner self-report, SMS/WhatsApp of a picture of the used HIVSS sent by partner or index, return of a used self-test to the facility by either the index or partner, and/or partner coming into facility for with an invitation for confirmatory testing or SOC counseling referral c. % of male partners with a positive HIV screening/test result d. % of newly diagnosed male partners who initiate ART within 3 months of diagnosis e. % of those on ART with viral suppression after 6 months on ART (index and partners)
3. In the intervention arm, we will assess acceptability and barriers (including safety/IPV) related to HIVSS distribution or use via surveys with all intervention participants who return for the study endline survey and a convenience samples of n=20 male partners (n=10 men who used HIVSS and n=10 men who did not use HIVSS)

ELIGIBILITY:
Inclusion Criteria:

1. Adult female 18+ years old
2. confirmed HIV-positive or on ART
3. confirmed to currently have a male partner and are sexually active
4. male partner is of HIV- or unknown status
5. confirmed to have a cell phone that can read and respond to SMS/WhatsApp messages
6. confirmed to be able to consent to study participation (no language constraints or psychological issues that would make it difficult to consent to participate in the study)

Exclusion Criteria:

Failure to meet all of inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2021-08-06 (Actual); Study Completion 2021-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Wall, PhD, Principal Investigator — Emory University; Kathryn Dovel, PhD, Study Director — University of California, Los Angeles; Dhirisha Naidoo, Study Director — BroadReach Healthcare
Locations (1):
- Department of Health Clinics, Nkangala, Mpumalanga, South Africa

IPD SHARING:
Plan to Share IPD: Undecided
Will be made available upon request to study team

REFERENCES:
- [Derived] Joseph Davey DL, Wall KM, Naidoo N, Naidoo D, Xaba G, Serao C, Malone T, Dovel K. HIV testing and linkage to ART following secondary distribution of HIV self-test kits to male partners of women living with HIV: a pilot randomized control trial in Mpumalanga, South Africa. J Int AIDS Soc. 2022 Jun;25(6):e25937. doi: 10.1002/jia2.25937. PMID 35690880

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HIV Self Testing | Standard of Care
Started | 86 | 94
Completed | 85 | 91
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIV Self Testing | Standard of Care | Total
Number analyzed (Participants) | 86 | 94 | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 86 | 94 | 180
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (8.6) | 36 (8.5) | 35 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 94 | 180
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 86 | 94 | 180
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 86 | 94 | 180

OUTCOME MEASURES:

1. Primary Outcome: Partner HIV Testing
Description: proportion of index partners who report testing
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Self Testing | Standard of Care
Number analyzed (Participants) | 86 | 91
Participants | 66 | 50
Statistical Analysis 1: Comparison: Standard of Care; Test type: Superiority; p < 0.05, Regression, Logistic; Risk Ratio (RR) = 1.41, 95% CI 2-sided [1.14 to 1.75]

2. Secondary Outcome: Positivity
Description: Proportion of male partners tested who test HIV+
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Self Testing | Standard of Care
Number analyzed (Participants) | 85 | 91
Participants | 9 | 6

3. Secondary Outcome: ART Initiation
Description: Proportion of male partners tested who initiate antiretroviral therapy (ART)
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Self Testing | Standard of Care
Number analyzed (Participants) | 9 | 6
Participants | 6 | 6

4. Secondary Outcome: Viral Suppression
Description: Proportion of male partners and index partners who achieve viral suppression
Time Frame: 3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From baseline to endline in the study (3 months)
Description: Any medical, social adverse event per DAIDS criteria
Arm/Group | HIV Self Testing | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/91
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/91
Other Adverse Events (participants affected / at risk) | 0/86 | 0/91

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/51/NCT05074251/Prot_SAP_ICF_000.pdf